CLINICAL TRIAL: NCT06191523
Title: The Effect of Melatonin as an Adjuvant Therapy for Preterm Neonates With Sepsis (Review of Malondialdehyde, Interleukin-6, Interleukin-8, Absolute Neutrophil Counts, and Sepsis Score)
Brief Title: The Effect of Melatonin as an Adjuvant Therapy for Preterm Neonates With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Sebelas Maret (Other)
Responsible Party: Principal Investigator, Dwi Hidayah, Doctoral Program, Universitas Sebelas Maret
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1.657/XII/HREC/2022
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Sepsis Newborn
Keywords: melatonin; sepsis; preterm neonates
MeSH Terms: conditions — Neonatal Sepsis; Sepsis | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): The control group will receive standard therapy and placebo.
  Interventions: Other: Control Group; Drug: Treatment Group
- Treatment Group (Experimental): The participants in the treatment group will receive standard therapy and a single dose of oral melatonin 20 mg
  Interventions: Other: Control Group; Drug: Treatment Group

INTERVENTIONS:
Other: Control Group — The control group will receive standard therapy and placebo.
Drug: Treatment Group — The participants in the treatment group will receive standard therapy and a single dose of oral melatonin 20 mg

SUMMARY:
The goal of this clinical trial is to assess the effect of melatonin on MDA serum, IL-6, IL-8 levels, ANC, and sepsis score in preterm neonates with sepsis. The main question aim to answer :

• Does melatonin affect MDA serum, IL-6, IL-8 levels, ANC, and sepsis score in preterm neonates with sepsis?

The participants in the treatment group will receive a single dose of oral melatonin 20 mg, meanwhile those the control group will receive placebo.

The researchers will compare MDA serum, IL-6, IL-8 levels, ANC, and sepsis score before and after receiving melatonin, whether there are decreases of MDA serum, IL-6, IL-8 levels, ANC and increase of sepsis score

ELIGIBILITY:
Inclusion Criteria:

* Newborns with gestational age of 28-36+6 weeks, birth weight according to gestational age, and diagnosis of sepsis based on HPS and PRS sepsis score criteria

Exclusion Criteria:

* Major congenital anomalies of the gastrointestinal tract.
* Continuous vomiting.
* Newborns with hypoxic ischemic encephalopathy (HIE), intracranial hemorrhage, feeding intolerance, necrotizing enterocolitis (NEC) and hormonal disorders.
* Septic shock.

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2023-04-27 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-Related Improvement of Sepsis Score Based on Gitto Scoring System | From enrollment to the end of treatment at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dwi Hidayah, Surakarta, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Henderson R, Kim S, Lee E. Use of melatonin as adjunctive therapy in neonatal sepsis: A systematic review and meta-analysis. Complement Ther Med. 2018 Aug;39:131-136. doi: 10.1016/j.ctim.2018.06.002. Epub 2018 Jun 11. PMID 30012383
- [Result] Gitto E, Karbownik M, Reiter RJ, Tan DX, Cuzzocrea S, Chiurazzi P, Cordaro S, Corona G, Trimarchi G, Barberi I. Effects of melatonin treatment in septic newborns. Pediatr Res. 2001 Dec;50(6):756-60. doi: 10.1203/00006450-200112000-00021. PMID 11726736
- [Result] El-Gendy FM, El-Hawy MA, Hassan MG. Beneficial effect of melatonin in the treatment of neonatal sepsis. J Matern Fetal Neonatal Med. 2018 Sep;31(17):2299-2303. doi: 10.1080/14767058.2017.1342794. Epub 2017 Jul 6. PMID 28612668
- [Result] El Frargy M, El-Sharkawy HM, Attia GF. Use of melatonin as an adjuvant therapy in neonatal sepsis. J Neonatal Perinatal Med. 2015;8(3):227-32. doi: 10.3233/NPM-15814072. PMID 26485549